### Administrative information:

| Sponsor name | Department of Infectious Diseases, Oslo University Hospital |
|---|---|
| Sponsor address | Oslo, Norway |
| EudraCT number / REC no | EudraCT number: 2014-004986-26 |
| Trial title | Therapeutic vaccination and immune modulation – new treatment strategies for the multidrug-resistant tuberculosis pandemic. An open label phase I clinical trial of the therapeutic TB H56:IC31 Vaccine and cyclooxygenase-inhibitors. |
| Trial ID | TBCOX2 |
| Trial registration number | ClinicalTrials.gov: NCT02503839 |

### SAP and protocol version:

| SAP version and date: | This SAP is version 1.0, dated 16.03.2020 |
|---|---|
| Protocol version | This document has been written based on information contained in the study protocol version 6.0, dated 12 October 2016 |

### **SAP** revision history:

| Protocol<br>version | SAP<br>version | Section number changed | Description and reason for change | Date changed |
|---|---|---|---|---|

Version Number: 1.0 Version Date: 16.03.2020 Corina Rueegg Oslo University Hospital 

### **SIGNATURE PAGE**

### PRINCIPAL/COORDINATING INVESTIGATOR:

Anne Ma Dyrhol-Riise, Professor Department of Infectious Diseases Oslo University Hospital

Signature 19/3 - 2020
Date (dd/mmm/yyyy)

#### TRIAL STATISTICIAN:

Corina S. Rueegg, PhD
Oslo Centre for Biostatistics and Epidemiology
Research Support Services
Oslo University Hospital

Signature 16.03.2020

Date (dd/mmm/yyyy)

### QC STATISTICIAN:

Inge Christoffer Olsen, PhD Clinical Trials Unit Research Support Services Oslo University Hospital

17/mar/2020

Date (dd/mmm/yyyy)

### **ABBREVIATIONS**

| AE | Adverse Event |
|--------|-----------------------------------------------|
| BCG | Bacille Calmette-Guérin |
| ВМІ | Body mass index |
| CI | Confidence Interval |
| COX-2i | COX-2 inhibitor |
| DMC | Data Monitoring Committee |
| eCRF | electronic Case Report Form |
| EAE | Expected Adverse Events (EAE) |
| ЕРТВ | Extra-pulmonary Tuberculosis |
| ESR | Erythrocyte Sedimentation Rate |
| Hb | Haemoglobin |
| ICS | Intracellular Cytokine Staining |
| IQR | Interquartile range |
| MDR-TB | Multidrug-Resistant Tuberculosis |
| MedDRA | Medical Dictionary for Regulatory Activities |
| QFT | Quantiferon |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| ТВ | Tuberculosis |
| WB | Whole Blood |
| XDR-TB | Extensively Drug-resistant Tuberculosis |

# **TABLE OF CONTENTS**

| 1 | INTRODUCTION | 5 |
|-----|-----------------------------------------------------------------|------|
| 201 | 1.1 Background and rationale | 5 |
| | 1.2 Trial Objectives | 5 |
| 2 | TRIAL METHODS | b |
| | 2.1 Trial Design | 6 |
| | 2.2 Randomisation | |
| | 2.3 Sample size | |
| | 2.4 Statistical Framework | 8 |
| | 2.5 Statistical Interim Analyses and Stopping Guidance | 12 |
| | 2.6 Timing of Final Analysis | 12 |
| | 2.7 Timing of Outcome Assessments | |
| 3 | STATISTIČAI PRINCIPLES | 13 |
| • | 3.1 Confidence Intervals and p-values | 13 |
| | 3.2 Adherence and Protocol Deviations | 13 |
| | 3.3 Analysis Ponulations | 15 |
| 4 | TRIAL POPULATION | |
| • | 4.1 Screening Data Fligibility, Recruitment, Withdrawal/Follow- | Jp15 |
| | 4.2 Raseline Patient Characteristics | 16 |
| 5 | ANALYSIS | 19 |
| • | 5.1 Outcome Definitions | 19 |
| | 5.2 Analysis Methods | 26 |
| 6 | S SAFETY ANALYSES | |
| 7 | Z STATISTICAL SOFTWARE | Zö |
| 8 | PEFERENCES | 28 |
| U | 8.1 Literature References | 28 |
| | 9.2 Reference to Data Handling Plan | 28 |
| Δ | ADDENDIX I _ THE CONSORT FLOW DIAGRAM | |
| | APPENDIX II – DATA HANDLINGS PLAN | 30 |

### 1 Introduction

This statistical analysis plan (SAP) is based on the guidelines for the content of SAPs in clinical trials<sup>1</sup> The SAP describes in detail the analyses to be conducted and highlights any deviations from the analysis described in the protocol. Deviations from methods described in the SAP, if any, will be specified in the clinical trial report. Reporting of the trial will take place after the data base lock.

# 1.1 Background and rationale

The World Health Organization estimates that globally 10.0 million people fell ill with active tuberculosis (TB) in 2018<sup>2</sup>. Globally, 3.4% of new TB cases and 18% of previously treated cases had multi-drugresistant TB (MDR-TB) which may take years to treat with expensive and toxic second-line drugs with uncertain efficacy. Further, the shifting of the TB epidemic towards extensively drug resistant (XDR-TB) with very restricted treatment options could reverse many of the major gains made in TB control and increase spread, morbidity and mortality. This calls for new treatment modalities, including host-directed therapy (HDT), that could be affordable and simple alternatives for a substantial number of patients with MDR-TB and XDR-TB in resource-poor countries.

# 1.2 Trial Objectives

### 1.2.1 Primary Objective

To evaluate the safety and tolerability of etoricoxib (Arcoxia) and the therapeutic TB vaccine H56:IC31 <u>alone and in combination</u> in patients with active TB disease treated with conventional 26-week anti-TB therapy.

### 1.2.2 Secondary Objectives

- a) To evaluate the effect of i) etoricoxib (Arcoxia) and ii) the therapeutic TB vaccine H56:IC31 on immunogenicity in patients with active TB disease treated with conventional 26-weeks anti-TB therapy. The immunogenicity endpoints are described and ranked according to importance in the sections 2.4.1 and 2.4.2 (Tables 1 and 2)
- b) To evaluate whether Arcoxia will improve the H56:IC31 TB vaccine response compared to H56:IC31 alone in patients with active TB disease treated with conventional 26-weeks anti-TB therapy. The H56:IC31 response endpoints are described and ranked according to importance in the sections 2.4.3 (Table 3)

### 1.2.3 Hypotheses

- 1. Etoricoxib administered during the first 84 days of 26-weeks standard TB treatment improves *Mycobacterium tuberculosis* (Mtb) specific immunity in patients with active TB disease (Comparison 1, **Figure 1**).
- 2. H56:IC31 vaccine administered at 2 doses (day 84 and day 140) during 26-weeks standard TB treatment induces H56:IC31 vaccine responses in patients with active TB disease (Comparison 2, Figure 1).

3. Etoricoxib administered during the first 140 days improves H56:IC31 vaccine responses in patients with active TB disease who are given the H56:IC31 vaccine administered at 2 doses (day 84 and day 140) during 26-weeks standard TB treatment (Comparison 3, Figure 1).



Figure 1: Illustration of the comparisons for each of the study hypotheses

### 2 Trial Methods

### 2.1 Trial Design

The TBCOX2 study is a randomized, open label, controlled, parallel group, multi-center, safety and explorative phase I study (**Figure 2**). The final treatment allocation to the four study arms is a 1:1:1:1 ratio with a randomization allocation ratio of first 2:2:1:0 for Group A and a subsequent randomization allocation ratio of 0:0:1:2 for Group B (see section 2.2 Randomization). Patients are randomized to either etoricoxib (COX-2 inhibitor (COX-2i); Arm 1 Arcoxia), TB vaccine (H56:IC31; Arm 2 H56:IC31), etoricoxib and TB vaccine (Arm 4 Arcoxia+H56:IC31), or no additional treatment (control arm; Arm 3 controls; **Figure 2**). In addition to these study-specific treatments, all study arms receive standard anti-TB therapy for 26 weeks (182 days), or longer in settings of single-drug resistance, drug intolerance or inadequate treatment response, as recommended by WHO treatment guidelines.

The study consists of two parts: The study starts with **Group A** that consists of full Arm 1, full Arm 2 and half of the control Arm 3. When safety data are satisfactory for all Group A participants at the safety interim analyses at study Day 98, **Group B** is enrolled and starting the study. Group B consists of half of the control Arm 3 and full Arm 4.



Figure 2: Study design of the TBCOX2 trial

### Treatments/Intervention

All patients receive standard anti-TB therapy for 26 weeks (day 0-182).

Add-on treatment will be given according to allocation:

Arm 1 (Arcoxia, target n=10): etoricoxib started at day 0 and given for 20 weeks (day 0-140)

Arm 2 (H56:IC31, target n=10): H56:IC31 vaccine administrated at day 84 and day 140.

Arm 3 (controls, target n=10): No add-on treatment.

Arm 4 (Arcoxia + H56:IC31, target n=10): etoricoxib started at day 0 and given for 20 weeks (day 0-140), H56:IC31 TB vaccine administrated at day 84 and day 140.

### Study groups

**Group A:** All patients allocated to Arm 1 (Arcoxia) and Arm 2 (H56:IC31). In addition, half of the patients allocated to Arm 3 (controls)

**Group B:** The other half of the patients allocated to Arm 3 (controls) and all patients allocated to Arm 4 (Arcoxia + H56:IC31)

### 2.2 Randomisation

By open label randomization TB patients meeting the inclusion criteria were included 2:2:1 in the Arms 1, 2 and 3 for Group A of the trial. When the last patient has reached study day 98 (2 weeks after the 1st H56:IC31 vaccine immunization) and safety of the treatments is found acceptable, participants for the Arms 4 and 3 will be recruited and randomized 2:1.

### 2.3 Sample size

No sample size calculation was performed as this is a Phase I trial. TBCOX2 is the first of its kind; exploratory, open label phase I study. Primary data on safety and efficacy of COX2-i (Arcoxia) as well as the H56:IC31 vaccine in patients with active TB are non-existing.


Based on the results in non-TB patients, this study aimed at including 40 patients, 10 in each arm (25 participants in Group A and 15 in Group B).

#### 2.4 Statistical Framework

This is a phase 1 exploratory trial where different hypotheses with different outcome variables will be tested. The current SAP describes the general models/methods applied for the statistical analysis of the trial. These methods will be applied to a list of hypotheses and outcome variables as hierarchically defined in the Tables 1 to 3 and 6 to 9. We will describe deviations from the general methods for individual hypothesis and outcome variables, if applicable.

Tables 1 to 3 give an overview of all the outcome variables of primary and secondary priority as well as the respective hypotheses tests and their hierarchical order for the interpretation of the results. Tables 6 to 9 define all the outcome variables generated (calculated and coded) within this SAP. Outcome variables that are listed in Tables 6-9 but not in Tables 1-3 are of tertiary priority.

### Explanation of outcomes described in Tables 1-3 and Tables 6-9:

- Sin cytokine: Cells expressing only one cytokine: sin\_IFNγ or sin\_IL2 or sin\_TNFα\*.
- Duo cytokine: Cells expressing two cytokines simultaneously: duo\_IFNγ/IL2 or duo\_IFNγ/TNFα\*or duo\_IL2/TNFα\*.
- Tri cytokines: Cells expressing three cytokines simultaneously: tri\_IFNγ/IL2/TNFα\*.
- Tot cytokines: SUM of cytokine combinations\_expressing cytokine of interest (sin\_cytokines PLUS duo\_cytokines PLUS tri\_cytokines\*): tot\_IFNγ or tot\_IL2 or tot\_TNFα\*
- All cytokines (CYTOKINE<sup>+</sup>) for Whole Blood ICS: SUM of the following cytokine combinations: tot\_IFNγ PLUS duo\_IL2/TNFα PLUS sin\_IL2 PLUS sin\_TNFα.
- All cytokines (CYTOKINE<sup>+</sup>) for Fluorospot: SUM of the following cytokine combinations: tot\_IFNγ PLUS tot\_IL2 MINUS duo\_IFNγ/IL2.

# Cytokine outcomes/responses as defined above are assessed by:

For the specific peptide stimulations: Ag85, ESAT6 (both 15aa, 10 overlapping peptide pools), CFP10 (25aa, 10, overlapping peptides), Rv2660 (20aa, 10 overlapping peptides). Purified Protein Derivate (PPD, 10μg/mL, SSI),

### Fluorospot (FS):

- SUM (Ag85+ESAT6): sum of respective cytokine response.
- SUM (Ag85+ESAT6+CFP10): sum of respective cytokine response.

#### Wholeblood (WB):

SUM (Ag85+ESAT6+Rv2660c) sum of respective cytokine response.

### 2.4.1 Outcome variables for Hypothesis 1

**Hypothesis 1:** Etoricoxib (Arcoxia) administered during the first 84 days of 26-weeks standard TB treatment improves Mtb specific immunity in patients with active TB disease

<sup>\*</sup> TNFa only for Whole Blood ICS.

Table 1: Hierarchal ranking of primary and secondary priority outcomes and definition of hypotheses that will be tested comparing Arcoxia vs. controls. Formal testing will be performed on the primary priority outcomes only, tertiary priority outcomes are not listed here.

| Method | Outcome | Time interval | Comparison |
|---|---|---|---|
| | Outcome | (days) | |
| Primary priority | | | |
| | All_cytokine responses to SUM | 0-84 | Arm (1+4) vs (2+3) |
| FILLODOCDOT /FC) | (Ag85+ESAT6+CFP10) | 0 04 | 7 (2 * 1) 00 (2 * 0) |
| FLUOROSPOT (FS) | Tot_IFNγ responses to SUM | 0-84 | Arm (1+4) vs (2+3) |
| | (Ag85+ESAT6+CFP10) | 0-04 | AIII (114) V3 (213) |
| Whole blood (WB) | All_cytokine CD4 responses to PPD | 0-84 | Arm (1+4) vs (2+3) |
| intracellular | All_cytokine CD4 responses to SUM | 0-84 | Arm (1+4) vs (2+3) |
| cytokine analyses | (Ag85+ESAT6+Rv2660) | 0-84 | AIII (114) V3 (213) |
| Secondary priority | | | |
| | All_cytokine responses to ESAT6 | 0-84 | Arm (1+4) vs (2+3) |
| | All_cytokine responses to Ag85 | 0-84 | Arm (1+4) vs (2+3) |
| FLUOROSPOT (FS) | All_cytokine responses to CFP10 | 0-84 | Arm (1+4) vs (2+3) |
| | Duo_IL2/IFNγ responses to SUM | 0-84 | Arm (1+4) vs (2+3) |
| | (Ag85+ESAT6+CFP10) | 0-84 | Aim (114) V3 (213) |
| | All_cytokine CD4/CD8 responses to | 0-84 | Arm (1+4) vs (2+3) |
| | ESAT6 | 0-04 | A(III (114) 43 (213) |
| | All_cytokine CD4/CD8 responses to | 0-84 | Arm (1+4) vs (2+3) |
| | Ag85 | 0-04 | 74111 (2:1) 43 (2:3) |
| | All_cytokine CD4/CD8 responses to | 0-84 | Arm (1+4) vs (2+3 |
| | Rv2660 | 0 5-1 | 7 (2 - 1, 12 (2 - 2, |
| Whole blood (WB) | Tri_IFNγ/IL2/TNFα CD4 responses to | 0-84 | Arm (1+4) vs (2+3) |
| intracellular | PPD | | |
| cytokine analyses | Tri_IFNγ/IL2/TNFα CD4 responses to | 0-84 | Arm (1+4) vs (2+3) |
| Cytokine analyses | SUM (Ag85+ESAT6+Rv2660) | | |
| | Duo_IL2/IFNγ CD4 responses to SUM | 0-84 | Arm (1+4) vs (2+3) |
| | (Ag85+ESAT6+Rv2660) | | |
| | Duo_IL2/IFNγ CD4 responses to PPD | 0-84 | Arm (1+4) vs (2+3) |
| | All_cytokines CD8 responses to PPD | 0-84 | Arm (1+4) vs (2+3) |
| | All_ cytokines CD8 responses to SUM | 0-84 | Arm (1+4) vs (2+3) |
| | (Ag85+ESAT6+Rv2660) | | |

### 2.4.2 Outcome variables for Hypothesis 2

**Hypothesis 2:** H56:IC31 vaccine administered at 2 doses (day 84 and day 140) during 26-weeks standard TB treatment induces H56:IC31 vaccine responses in patients with active TB disease.

Table 2: Hierarchal ranking of primary and secondary priority outcomes and definition of hypotheses that will be tested comparing H56:IC31 vs. controls. Formal testing will be performed on the primary priority outcomes only, tertiary priority outcomes are not listed.

| Method | Outcome | Time interval<br>(days) | Comparison |
|---|---|---|---|
| Primary priority | | | |
| | All_cytokine responses to H56 | 84-154 | Arm 2 vs 3 |
| FILLODOSDOT /FS) | Tot_IFNγ responses to H56 | 84-154 | Arm 2 vs 3 |
| FLUOROSPOT (FS) | All_cytokine responses to SUM (Ag85+ESAT6) | 84-154 | Arm 2 vs 3 |
| Whole blood (WB) intracellular cytokine analyses | All_cytokine CD4 responses to SUM (Ag85+ESAT6+Rv2660) | 84-154 | Arm 2 vs 3 |
| Serology/antibody measurements | IgG antibody responses to H56: IC31 | 84-154 | Arm 2 vs 3 |
| Secondary priority | | · | • |
| | All_cytokine responses to ESAT6 | 84-154 | Arm 2 vs 3 |
| | All_cytokine responses to Ag85 | 84-154 | Arm 2 vs 3 |
| | All_cytokine responses to CFP10 | 84-154 | Arm 2 vs 3 |
| FILLODOCDOT (FC) | Duo_IL2/IFNγ responses to H56 | 84-154 | Arm 2 vs 3 |
| FLUOROSPOT (FS) | Tot_IFNγ responses to SUM (Ag85+ESAT6) | 84-154 | Arm 2 vs 3 |
| | Duo_IL2/IFNγ responses to SUM (Ag85+ESAT6) | 84-154 | Arm 2 vs 3 |
| | All_cytokine CD4/CD8 responses to ESAT6 | 84-154 | Arm 2 vs 3 |
| | All_cytokine CD4/CD8 responses to Ag85 | 84-154 | Arm 2 vs 3 |
| | All_cytokine CD4/CD8 responses to Rv2660 | 84-154 | Arm 2 vs 3 |
| Whole blood (WB) intracellular | All_cytokine CD4/CD8 responses to PPD | 84-154 | Arm 2 vs 3 |
| cytokine analyses | Tri_IFNy/IL2/TNFα CD4 responses to SUM (Ag85+ESAT6+Rv2660) | 84-154 | Arm 2 vs 3 |
| | Duo_IL2/IFNγ CD4 responses to SUM (Ag85+ESAT6+Rv2660) | 84-154 | Arm 2 vs 3 |
| | All_cytokine CD8 responses to SUM (Ag85+ESAT6+Rv2660) | 84-154 | Arm 2 vs 3 |

### 2.4.3 Outcome variables for Hypothesis 3

**Hypthesis 3:** Etoricoxib (Arcoxia) administered during the first 140 days of 26-weeks standard TB treatment improves H56:IC31 vaccine responses given at 2 doses (day 84 and day 140) in patients with active TB disease.


Table 3: Hierarchal ranking of primary and secondary priority outcomes and definition of hypotheses that will be tested comparing Arcoxia + H56:IC31 vs. H56:IC31 alone. Formal testing will be performed on the primary priority outcomes only, tertiary priority outcomes are not listed.

| Method | Outcome | Time interval<br>(days) | Comparison |
|---|---|---|---|
| Primary priority | | | |
| | All_cytokine responses to H56 | 84-154 | Arm 4 vs 2 |
| | Tot_IFNγ responses to H56 | 84-154 | Arm 4 vs 2 |
| FLUOROSPOT (FS) | All_cytokine responses to SUM (Ag85+ESAT6) | 84-154 | Arm 4 vs 2 |
| Whole blood (WB) intracellular cytokine analyses | All_cytokine CD4 responses to SUM (Ag85+ESAT6+Rv2660) | 84-154 | Arm 4 vs 2 |
| Serology/antibody<br>measurements | IgG antibody responses to H56:IC31 | 84-154 | Arm 4 vs 2 |
| Secondary priority | | | |
| | All_cytokine responses to ESAT6 | 84-154 | Arm 4 vs 2 |
| | All_cytokine responses to Ag85 | 84-154 | Arm 4 vs 2 |
| | All_cytokine responses to CFP10 | 84-154 | Arm 4 vs 2 |
| | Duo_IL2/IFNγ responses to H56 | 84-154 | Arm 4 vs 2 |
| FLUOROSPOT (FS) | Tot_IFNγ FS responses to SUM (Ag85+ESAT6) | 84-154 | Arm 4 vs 2 |
| | Duo_IL2/IFNγ FS responses to SUM (Ag85+ESAT6) | 84-154 | Arm 4 vs 2 |
| | All_cytokine CD4/CD8 responses to ESAT6 | 84-154 | Arm 4 vs 2 |
| | All_cytokine CD4/CD8 responses to Ag85 | 84-154 | Arm 4 vs 2 |
| | All_cytokine CD4/CD8 responses to Rv2660 | 84-154 | Arm 4 vs 2 |
| Whole blood (WB) intracellular | All_cytokine CD4/CD8 responses to PPD | 84-154 | Arm 4 vs 2 |
| cytokine analyses | Tri_IFNγ/IL2/TNFα CD4 responses to SUM (Ag85+ESAT6+Rv2660) | 84-154 | Arm 4 vs 2 |
| | Duo_IL2/IFNγ CD4 responses to SUM (Ag85+ESAT6+Rv2660) | 84-154 | Arm 4 vs 2 |
| | All_cytokine CD8 responses to SUM (Ag85+ESAT6+Rv2660) | 84-154 | Arm 4 vs 2 |

### 2.4.4 Hypothesis Test

This study is an exploratory, hypothesis generating phase I trial. There will be no formal statistical hypotheses testing as part of the analyses of this trial. All group comparisons including p-values will be hypothesis supporting and not interpreted as confirmatory. Because of the exploratory nature of

the trial, there will be no adjustment for multiple testing. The importance of the interpretation of the statistical test/results is defined by the hierarchical ranking in Tables 1 to 3. An increase in immune response will be interpreted as the favourable outcome.

#### 2.4.5 Decision Rule

Group comparisons resulting in a p-value below 0.05 will be denoted as a statistically significant difference, but no claim of superiority either way will be made based on such findings.

# 2.5 Statistical Interim Analyses and Stopping Guidance

There will be no efficacy interim analyses in this trial. The safety of etoricoxib and H56:IC31 was determined when all participants of Group A reached day 98. After the approval of the safety, the enrolment into arm 4 was started.

# 2.6 Timing of Final Analysis

When all participants have reached day 238.

### 2.7 Timing of Outcome Assessments

**Table 4. Study flow chart** gives an overview of the outcomes assessed at the different time points in the study. The detailed methods of all procedures are described in the protocol chapter 10.4.

| | | | Folle | End of study | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study day | Screen | 0 | 7 | 14 | 28 | 56 | 84 | 98 | 140 | 154 | 182 | 210 | 238 |
| Window (days) | | NA | ±2 | ±2 | ±7 | ±7 | <b>±</b> 7 | 23 | ±7 | ±3 | ±7 | ±14 | ±14 |
| Informed consent | х | | | | | | | | | | | | |
| Inclusion/exclusion<br>evaluation | х | | | | | | | | | | | | |
| Demographics/<br>medical history | Х | | | | | | | | | | | | ļ.,, |
| AFS/Culture/Xpert <sup>()</sup> | Х | X | | X* | | X* | X | | Х | | X | | Х |
| Radiology <sup>2)</sup> | х | | | | | Х | | | | | X | | |
| TB chemotherapy <sup>3)</sup> | | Х | X | X | Х | Х | Х | X | X | X | Х | | |
| Physical<br>Examination <sup>4)</sup> | х | х | × | X | Х | Х | Х | Х | X | Х | X | х | X |
| Vital signs <sup>5)</sup> | х | Х | X | х | X | Х | Х | Х | X | X | X | Х | X |
| Symptoms (6) | х | х | Х | Х | х | X | Х | × | Х | X | X | Х | X |
| Treatment<br>(etoricoxib) | | Х | х | х | Х | Х | Х | Х | X | | | | |
| Haematology/clinical chemistry <sup>6)</sup> | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | X | X | X |
| Pharmacokinetics <sup>7)</sup> | | | X | | | | | | | | | | |
| Adverse events | | | Х | х | Х | Х | X | X | X | X | X | X | X |
| Con. Medication | X | Х | Х | х | X | X | X | X | X | X | X | Х | X |
| Vaccine adm. (T) <sup>8)</sup> | | | | | | | т | | T | | | | |
| Blood sampling for exploratory ssays | | X | | х | х | х | х | х | х | х | X | X | X |
| Vaccine IgG <sup>9)</sup> | | X | | | | | X | X | X | X | | | X |
| RNA analysis <sup>9)</sup> | | X | | | | | х | х | X | х | | | X |
| PBMC ICS® | | x | | | | | X | X | X | X | | | X |

<sup>1).</sup> AFS, cubuse, microscopy, PCR/GeneXpert as part of routine clinical evaluation of TB. 2) Appropriate radiology (ches) X-ray-CTA/(RNUL/PET) taken as part of clinical evaluation × E-morth settore entering the study. 3) Arth-TB chemotherapy; standard combination by make day 0-56, continuation phase day 0-56, continuation phase day 56-162. 6) Physical examination by clinical investigator at every visit, the eatent depending on the chircal situation in the case of glanduatr TB, the clancy(s) are measured. 5) Blood pressure, pulse, temperature. 6) Hb, Lpk, monocytes, symphocytes, symphocytes, pymphocytes, Tpk, ESR, CRP, SR, Na, K, Ca, creatione, ASAT, ALAT, LDH, bdrubin, armylase, CK, croatstend, glucose, gGT, urine acid, 5-oCG) at every visit. OFT-TB at day 0 and 182, 7). Study

# 3 Statistical Principles

# 3.1 Confidence Intervals and p-values

All calculated p-values will be two-sided and compared to a 5% significance level. If a p-value is less than 0.05, the corresponding group difference will be denoted as statistically significant. All estimates will be presented with two-sided 95% confidence intervals.

### 3.2 Adherence and Protocol Deviations

### 3.2.1 Adherence to Allocated Treatment

All subjects who have received at least one dose of etoricoxib (Arcoxia) and/or H56:IC31-vaccine are included in the safety analysis. Because of the hypothesis generating nature of the trial (phase I) no subjects will be excluded from the analysis because of lack of adherence.

Below are the definitions of treatment adherence. If the following conditions are reached, a person is considered compliant:

All arms: No corticosteroids/ additional NSAIDs the last 7 days prior to biobank sampling for immunogenicity read-outs.

### Additional requirements for the specific treatment arms:

Arm 1, allocated to etoricoxib treatment: during the intervention period (Day 0-140), ≥80% of the expected number of tablets were taken. Number of tablets taken was recorded by asking the participants and having them return the pill container.

Arm 2 allocated to H56:IC31-vaccine: having received ≥1 dose(s) of the H56:IC31-vaccine.

Arm 4 allocated to etoricoxib treatment and H56:IC31-vaccine: 1) during the intervention period (Day 0-140), ≥80% of the expected number of tablets were taken; AND, 2) having received ≥1 dose(s) of the H56:IC31-vaccine. Number of tablets taken was recorded by asking the participants and having them returned the pill container.

The number (and percentage) of patients that were compliant will be summarised by treatment group with details for reasons of non-compliance. The results will be shown for the Randomised Set, Safety Analysis Set and Full Analysis Set (see Section 3.3. Analysis Populations). No formal statistical testing will be undertaken.

#### 3.2.2 Protocol Deviations

The following are pre-defined major protocol deviations. The protocol deviations will be described in the article:

- Entering the trial when the eligibility criteria should have prevented trial entry
- Discontinuation of intervention, thus not adhering to the allocated treatment as described in 3.2.1.
- Use of sporadic COX-inhibitor/NSAIDS not according the allocated treatment as described in 3.2.1.
- Received or used a different intervention than the one allocated to.

The number (and percentage) of patients with major protocol deviations will be summarised by treatment group with details of type of deviation provided. The results will be shown for the Randomised Set, Safety Analysis Set and Full Analysis Set (see Section 3.3. Analysis Populations). No formal statistical testing will be undertaken.

### 3.3 Analysis Populations

#### **Enrolled Set:**

All patients who have provided informed consent and have been entered into the study database.

#### **Randomised Set:**

All patients randomly assigned to a treatment group.

#### Safety Analysis Set (SAS):

All patients of the randomised set having received at least one dose of the allocated treatment (meaning no treatment for the controls and the first phase of the vaccination arm). Subjects who withdrew from the study due to own wish to discontinue his/her participation in the study were not followed-up and no safety information after withdrawal is available. The patient will still be followed and receive standard anti-TB chemotherapy for 26 weeks or as long as needed as determined by the responsible clinician according to clinical guidelines. A list of withdrawn subjects, with the reasons for withdrawal, will be presented in the article. Participants are included in the safety analysis until loss to follow-up or end of study, whatever comes first. Any significant AE will be followed-up by the responsible clinician according to clinical guidelines until the AE is resolved.

The safety analysis will be divided into AE/SAE happening within the following three time periods:

- a. Day 0 to day 84 (or date of first vaccination if applicable).
- b. Day 85 (or date of first vaccination if applicable) to day 154 (or 14 days after last vaccination/last Arcoxia treatment, if applicable).
- c. Day 155 (or 15 days after last vaccination/last Arcoxia treatment, if applicable) to day 238.

If the second vaccination is missing, day 154 is defined as 70 days after the date of day 84.

#### Full Analysis Set (FAS):

All patients of the randomised set with at least one valid measurement of any of the outcome variables listed in Tables 6-9. We will perform intention to treat (ITT) analysis in the FAS, meaning that we treat participants as they were randomized and independent of adherence. Per protocol analyses will not be performed because of the generally good adherence observed by the study group.

# 4 Trial Population

# 4.1 Screening Data, Eligibility, Recruitment, Withdrawal/Follow-up

The total number of screened patients and reasons for not entering the trial will be summarised and tabulated.

A CONSORT flow diagram (Appendix I) will be used to summarise the number of patients who were:

- screened and not eligible
- screened and eligible
- eligible and randomised (corresponding to the Randomised Set)
- eligible but not randomised\*
- received the randomised allocation (corresponding to Safety Analysis Set)

- did not receive the randomised allocation\*
- lost to follow-up\*
- discontinued the intervention\*
- withdrew consent\*
- randomised and included in the primary analysis (corresponding to Full Analysis Set)
- randomised and excluded from the primary analysis\*
- completers

### 4.2 Baseline Patient Characteristics

The following patient demographics and baseline characteristics will be summarised (example Table 5): gender (male, female), age, ethnicity (Caucasian, Black, Asian, other), smoking (yes, no, unknown), alcohol use >3units/week (yes, no, unknown), drug abuse (yes, no, unknown), Bacille Calmette-Guérin (BCG) vaccine scar (yes, no), co-morbidities (allergy, kidney failure, previous gastric ulcer/GI bleeding, liver disease/failure, chronic pulmonary disease, other medical condition), previous TB treatment (yes, no), TB diagnosis (pulmonary, pulmonary/extrapulmonary), Extrapulmonary location (no EPTB, lymphadenitis, bone/joint/soft tissue, pleuritis, abdominal, urogenital, other), radiology (infiltrate, cavity, miliary, pleural fluid, mediastinal changes, extrapulmonary), symptoms of cough, chest pain, night sweat with grading 0-5 (no symptoms, 1 symptom, ≥2 symptoms), QFT result (positive, intermediate, negative), vital signs [weight (kg), BMI (kg/m²), body temperature (°Celsius)], and laboratory parameters (haemoglobin (Hb), Erythrocyte Sedimentation Rate (ESR), CRP and Quantiferon-TB (QFT)).

Patient demographics and baseline characteristics will be summarised by randomised treatment arm and overall using descriptive statistics: median, interquartile range (IQR), minimum, and maximum for continuous variables, and number and percentages of patients for categorical variables. There will be no formal statistical testing of differences between the arms. Any clinical important imbalance between the treatment groups will be noted.

**Table 5** shows a table draft for the baseline patient characteristics to be displayed in the article. The Table will be presented for the FAS (Suppl. Appendix) and the SAS (in the Paper) separately.

<sup>\*</sup>reasons will be provided.

Table 5: Draft table of the baseline patient characteristics to be displayed in the article

| | Total<br>N= | | Arm 1<br>N= | | Arm 2<br>N= | | Arm 3<br>N= | | Arm 4<br>N= | |
|---|---|---|---|---|---|---|---|---|---|---|
| Categorical variables | N | % | N | % | N | % | N | % | N | % |
| Gender | | | | | | | | | | |
| Male | | | | | | | | | | |
| Female | | | | | | | | | | |
| Ethnicity | | | | | | | | | | |
| Caucasian | | | | | | | | | | |
| Black | | | | | | | | | | |
| Asian | | | | | | | | | | |
| Other | | | | | | | | | | |
| Smoking status | | | | | | | | | | |
| Yes | | | | | | | | | | |
| No | | | | | | | | | | |
| Unknown | | | | | | | | | | |
| Alcohol use >3 | | | | | | | | | | |
| units/week | | | | | | | | | | |
| Yes | | | | | | | | | | |
| No | | | | | | | | | | |
| Unknown | | | | | | | | | | |
| Drug abuse | | | | | | | | | | |
| Yes | | | | | | | | | | |
| No | | | | | | | | | | |
| Unknown | | | | | | | | | | |
| BCG scar | | | | | | | | | | |
| Yes | | | | | | | | | | |
| No | | | | | | | | | | |
| Co-morbidities <sup>a</sup> | | | | | | | | | | |
| Allergy | | | | | | | | | | |
| Kidney failure | | | | | | | | | | |
| Previous gastric | | | | | | | | | | |
| ulcer/GI bleeding | | | | | | | | | | |
| Liver disease | | | | | | | | | | |
| Chronic pulmonary | | | | | | | | | | |
| disease<br>Other medical | | | | | | | | | | |
| condition | | | | | | | | | | |
| Previous TB treatment | 11-11- | | | | | | | | | |
| Yes Yes | | | | | | | | | | |
| No | | | | | | | | | | |
| TB diagnosis | | | | | | | | | | |
| Pulmonary<br>Pulmonary/ | | | | | | | | | | |
| extrapulmonary | | | | | | | | | | |
| Extrapulmonary | | | | | | | | | | |


| Lymphadenitis<br>Bone/joints/soft tissue<br>Pleuritis<br>Abdominal<br>Urogenital<br>Other | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Radiology | | | | | | | | | | |
| Infiltrate | | | | | | | | | | |
| Cavity | | | | | | | | | | |
| Miliary | | | | | | | | | | |
| Pleural fluid | | | | | | | | | | |
| Mediastinal changes | | | | | | | | | | |
| Extrapulmonary | | | | | | | | | | |
| Symptoms (cough, chest | | | | | | | | | | |
| pain, night sweat) | | | | | | | | | | |
| No symptoms | | | | | | | | | | |
| 1 symptom | | | | | | | | | | |
| ≥2 symptoms | | | | | | | | | | |
| QFT result | | | | | | | | | | |
| Positive | | | | | | | | | | |
| Indeterminate | | | | | | | | | | |
| Negative | | | | | | | | | | |
| Continuous variables | | IQR | | IQR | | IQR | | IQR | B. A. a. di a. ua | IQR |
| | Median | (range) | Median | (range) | Median | (range) | Median | (range) | Median | (range) |
| Age (years) | | | | | | | | | | |
| Vital signs | | | | | | | | | | |
| Weight (kg) | | | | | | | | | | |
| BMI (kg/m²) | | | | | | | | | | |
| Body temperature (°C) | | | | | | | | | | |
| Hb (g/dl) | | | | | | | | | | |
| QFT (IU/ml) | | | | | | | | | | |
| ESR (mm) | | | | | | | | | | |
| CRP | | | | | | | | | | |

Abbreviations: BCG, Bacille Calmette-Guérin; BMI, body mass index; EPTB, extra-pulmonary Tuberculosis; ESR, Erythrocyte Sedimentation Rate; Hb, haemoglobin; IQR, interquartile range; N, number; QFT, Quantiferon. CRP, C-Reactive Protein.


<sup>&</sup>lt;sup>a</sup> Numbers and proportions of patients having the respective co-morbidity.

### 5 Analysis

#### 5.1 Outcome Definitions

### 5.1.1 General Definitions and Derived Variables

### 5.1.1.1 Baseline characteristics:

All baseline characteristics variables are listed and described in **Table 5** and section 4.2 Baseline Patient Characteristics.

There is only one derived variable among them:

 Body Mass Index (BMI) at baseline is calculated as follows from weight and height assessed at Screening visit/Day 0:

BMI=weight in kg/(height in m)2

### 5.1.1.2 Safety outcomes:

General definitions and derived variables for safety measurements are listed under 4.1.2 Primary Outcome Definition.

### 5.1.1.3 Immunogenicity read-outs:

The calculation and definition of the immunogenicity outcomes are described in Tables 6-9. The immunogenicity outcomes were generated by three analysis methods, briefly explained below:

- 1. FluoroSpot: FluoroSpot is a variation of the enzyme-linked immune absorbent spot (ELISpot) assay. It measures the number of thawed peripheral blood mononuclear cells (PBMC) secreting IFN-γ or IL-2 or both cytokines (spot forming units (SFC) per 300.000 PBMCs by adding 2 different fluorophore tags to the antibodies targeting IFN-γ (wavelength 250) and IL-2 (wavelength 630). For each time-point analysed per study subject, these repeated measurements are performed for each of 4 different stimulatory conditions (ESAT6, Ag85b, CFP10, H56) as well as a negative and a positive (CD3) control. The derived outcomes are defined in Table 6. The unit for all FluoroSpot outcomes is SFC/300.000 PBMC.
- 2. Whole-blood intracellular cytokine staining and flowcytometry (WB-ICS): Freshly drawn whole blood (WB) from study participants at each time-point was separated in aliquots with various stimulation (ESAT6, Ag85b, Rv2660c, PPD) prior to freezing and storage. Samples are then thawed, stained with fluorescent antibodies and analysed by flow cytometry characterizing phenotypic markers and cytokine production in CD4+ and CD4- (=CD8+) T cells. The derived outcomes are defined in Table 7 (CD4+) and Table 8 (CD8+).
- Serology analysis: IgG antibodies against the vaccine fusion protein H56:IC31 was analysed in singlets by enzyme-linked immunosorbent assay (ELISA). Variables are used as given in the dataset, no derived outcome variables or calculations. The serology outcomes are listed in Table 9.

Table 6: Definition of derived outcomes from the FluoroSpot (FS) analysis

| Outcome priority group | | | Derived outcome |
|---|---|---|---|
| Tertiary | tot_IFNγ (FS) | ESAT6 | Mean(triplicates ESAT6) – mean(triplicates negative control) |
| Tertiary | tot_IFNγ (FS) | Ag85 | Mean(triplicates Ag85) – mean(triplicates negative control) |
| Tertiary | tot_IFNγ (FS) | CFP10 | Mean(triplicates CFP10) – mean(triplicates negative control) |
| Primary H2²/H3³ | tot_IFNγ (FS) | H56 | Mean(triplicates H56) – mean(triplicates negative control) |
| Primary H1¹ | tot_IFNy (FS) | SUM (ESAT6+<br>Ag85+CFP10) | SUM of (tot_IFNy) for ESAT6, Ag85,CFP10 |
| Secondary H2 <sup>2</sup> /H3 <sup>3</sup> | tot_IFNγ (FS) | SUM (ESAT6+<br>Ag85) | SUM of (tot_IFNy) for ESAT6, Ag85 |
| Tertiary | tot_IL2 (FS) | ESAT6 | Mean(triplicates ESAT6) – mean(triplicates negative control) |
| Tertiary | tot_IL2 (FS) | Ag85 | Mean(triplicates Ag85) – mean(triplicates negative control) |
| Tertiary | tot_IL2 (FS) | CFP10 | Mean(triplicates CFP10) – mean(triplicates negative control) |
| Tertiary | tot_IL2 (FS) | H56 | Mean(triplicates H56) – mean(triplicates negative control) |
| Tertiary | Tot_IL2 (FS) | SUM (ESAT6+<br>Ag85+CFP10) | SUM of (tot_IL2) for ESAT6, Ag85 |
| Tertiary | Tot_IL2 (FS) | SUM (ESAT6+<br>Ag85) | SUM of (tot_IL2) for ESAT6, Ag85, CFP10 |
| Tertiary | duo_IFNγ/IL2 (FS) | ESAT6 | Mean(triplicates ESAT6) – mean(triplicates negative control) |
| Tertiary | duo_IFNγ/IL2 (FS) | Ag85 | Mean(triplicates Ag85) – mean(triplicates negative control) |
| Tertiary | duo_IFNγ/IL2 (FS) | CFP10 | Mean(triplicates CFP10) – mean(triplicates negative control) |
| Secondary H2 <sup>2</sup> /H3 <sup>3</sup> ,<br>Tertiary H <sup>1</sup> | duo_IFNy/IL2 (FS) | H56 | Mean(triplicates H56) – mean(triplicates negative control) |
| Secondary H <sup>1</sup> | duo_IFNy/IL2 (FS) | SUM (ESAT6+<br>Ag85+CFP10) | SUM of (duo_IFNy/IL2) for ESAT6, Ag85, CFP10 |
| Secondary H <sup>2</sup> /H <sup>3</sup> | duo_IFNy/IL2 (FS) | SUM ESAT6+<br>Ag85) | SUM of (duo_IFNy/IL2) for ESAT6, Ag85 |
| Secondary | all_ Cytokine (FS) | ESAT6 | tot_IFNy + tot_IL2 - duo_IFNy/IL2 for ESAT6 |
| Secondary | all_ Cytokine (FS) | Ag85 | tot_IFNy + tot_IL2 - duo_IFNy/IL2 for Ag85 |
| Secondary | all_ Cytokine (FS) | CFP10 | tot_IFNy + tot_IL2 - duo_IFNy/IL2 for CFP10 |
| Primary H2 <sup>2</sup> /H3 <sup>3</sup> | all_Cytokine (FS) | H56 | tot_IFNy + tot_IL2 - duo_IFNy/IL2 for H56 |
| Primary H2²/H3³ | all_Cytokine (FS) | SUM (ESAT6+<br>Ag85) | SUM of (tot_IFNy + tot_IL2 - duo_IFNy/IL2) for ESAT6, Ag85 |
| Primary H1 <sup>1</sup> | all_Cytokine (FS) | SUM (ESAT6+<br>Ag85+CFP10) | SUM of (tot_IFNy + tot_IL2 - duo_IFNy/IL2) for ESAT6, Ag85, CFP10 |

<sup>1</sup>Hypothesis 1 (etoricoxib). <sup>2</sup>Hypothesis 2 (H56:IC31 vaccine). <sup>3</sup>Hypothesis 3 (etoricoxib + H56:IC31 vaccine).

Note: For a valid IFN $\gamma$  result, the following conditions must be fulfilled: the SFU/SFC value (mean of duplicates) for IFN $\gamma$  at CD3 (positive control) is 1) >12 AND 2)  $\geq$ 2 times the SFU/SFC value (mean of triplets) for IFN $\gamma$  at the negative control.

**Colour code**: blue=secondary priority; red=primary priority; white=tertiary priority.

Table 7: Definition of derived outcomes from the *whole-blood* (WB) intracellular cytokine staining and flow cytometry analysis for CD4+ (eg. CD3+ CD4+ CD8-)\*

| Outcome<br>priority group | Immunology readout | Stimulation | Derived outcome |
|---|---|---|---|
| Tertiary | sin_IFNγ (WB) | ESAT6 | %(CD4+ESAT6) - %(CD4+ Unstim) |
| Tertiary | sin_IFNγ (WB) | Ag85 | %(CD4+ Ag85b) - %(CD4+ Unstim) |
| Tertiary | sin_IFNγ (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Tertiary | sin_IFNγ (WB) | PPD | %(CD4+ PPD) - %(CD4+ Unstim) |
| Tertiary | sin_IL2 (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim) |
| Tertiary | sin_IL2 (WB) | Ag85 | %(CD4+ Ag85b) – %(CD4+ Unstim) |
| Tertiary | sin_IL2 (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Tertiary | sin_IL2 (WB) | PPD | %(CD4+ PPD) – %(CD4+ Unstim) |
| Tertiary | sin_TNFα (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim) |
| Tertiary | sin_TNFα (WB) | Ag85 | %(CD4+ Ag85b) - %(CD4+ Unstim) |
| Tertiary | sin_TNFα (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Tertiary | sin_TNFα (WB) | PPD | %(CD4+ PPD) - %(CD4+ Unstim) |
| Tertiary | duo_IFNγ/IL2 (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim |
| Tertiary | duo_IFNγ/IL2 (WB) | Ag85 | %(CD4+ Ag85b) – %(CD4+ Unstim) |
| Tertiary | duo_IFNγ/IL2 (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Secondary H1 | duo_IFNγ/IL2 (WB) | PPD | %(CD4+ PPD) – %(CD4+ Unstim) |
| Tertiary | duo_IFNγ/TNFα (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim) |
| Tertiary | duo_IFNγ/TNFα (WB) | Ag85 | %(CD4+ Ag85b) - %(CD4+ Unstim) |
| Tertiary | duo_IFNγ/TNFα (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Tertiary | duo_IFNγ/TNFα (WB) | PPD | %(CD4+ PPD) - %(CD4+ Unstim) |
| Tertiary | duo_TNFα/IL2 (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim) |
| Tertiary | duo_TNFα/IL2 (WB) | Ag85 | %(CD4+ Ag85b) - %(CD4+ Unstim) |
| Tertiary | duo_TNFα/IL2 (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Tertiary | duo_TNFα/IL2 (WB) | PPD | %(CD4+ PPD) - %(CD4+ Unstim) |
| Tertiary | tri_IFN $\gamma$ /IL2/TNF $\alpha$ (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim) |
| Tertiary | tri_IFNγ/IL2/TNFα (WB) | Ag85 | %(CD4+ Ag85) - %(CD4+ Unstim) |
| Tertiary | $tri_IFN\gamma/IL2/TNF\alpha$ (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Secondary H1 | tri_IFNy/IL2/TNFα (WB) | PPD | %(CD4+ PPD) - %(CD4+ Unstim) |
| Tertiary | tot_IFNγ (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim) |
| Tertiary | tot_IFNγ (WB) | Ag85 | %(CD4+ Ag85) - %(CD4+ Unstim) |
| Tertiary | tot_IFNγ (WB) | Rv2660c | %(CD4+ RV2660c) - %( CD4+ Unstim) |
| Tertiary | tot_IFNγ (WB) | PPD | %(CD4+ PPD) - %(CD4+ Unstim) |
| Tertiary | tot_IFNγ (WB) | SEB* | %(CD4+ SEB) - %(CD4+ Unstim) |


| Tertiary | tot_IL2 (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim) |
|---|---|---|---|
| Tertiary | tot_IL2 (WB) | Ag85 | %(CD4+ Ag85) - %(CD4+ Unstim) |
| Tertiary | tot_IL2 (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Tertiary | tot_IL2 (WB) | PPD | %(CD4+ PPD) - %(CD4+ Unstim) |
| Tertiary | tot_TNFα (WB) | ESAT6 | %(CD4+ ESAT6) - %(CD4+ Unstim) |
| Tertiary | tot_TNFα (WB) | Ag85 | %(CD4+ Ag85) - %(CD4+ Unstim) |
| Tertiary | tot_TNFα (WB) | Rv2660c | %(CD4+ RV2660c) - %(CD4+ Unstim) |
| Tertiary | tot_TNFα (WB) | PPD | %(CD4+ PPD) - %(CD4+ Unstim) |
| Secondary | All_Cytokine WB | ESAT6 | SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 |
| Secondary | All_Cytokine WB | Ag85 | SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 |
| Secondary | All_Cytokine WB | Rv2660c | SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c |
| Primary H1 <sup>1</sup> ,<br>Secondary<br>H2 <sup>2</sup> /H3 <sup>3</sup> | All_Cytokine WB | PPD | SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD |
| Primary | All_Cytokine WB | SUM (ESAT6+<br>Ag85+Rv2660c) | SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6, Ag85 and Rv2660c |
| Secondary | tri_ cytokines (WB) | SUM (ESAT6+<br>Ag85+Rv2660c) | SUM of (tri_IFNγ/IL2/TNFα) for ESAT6, Ag85 and Rv2660c |
| Secondary | duo_IFNy/IL2 (WB) | SUM (ESAT6+<br>Ag85+Rv2660c) | SUM of (duo_IFNy/IL2) for ESAT6, Ag85 and Rv2660c |
| Tertiary | duo_IFNγ/TNFα (WB) | SUM (ESAT6+<br>Ag85+Rv2660c) | SUM of (duo_IFNγ/TNFα) for ESAT6, Ag85 and Rv2660c |
| Tertiary | duo_ IL2/TNFα/ (WB) | SUM (ESAT6+<br>Ag85+Rv2660c) | SUM of (duo_IL2/TNFα) for ESAT6, Ag85 and Rv2660c |

<sup>1</sup>Hypothesis 1 (etoricoxib). <sup>2</sup>Hypothesis 2 (H56:IC31 vaccine). <sup>3</sup>Hypothesis 3 (etoricoxib + H56:IC31 vaccine).

Colour code: blue=secondary priority; red=primary priority; white=tertiary priority.

Table 8: Definition of derived outcomes from the whole-blood (WB) intracellular cytokine staining and flow cytometry analysis for CD8+ (eg.CD3+ CD4- CD8+)

| Outcome<br>priority group | Immunology readout | Stimulation | Derived outcome |
|---|---|---|---|
| Tertiary | sin IFNγ (WB) | ESAT6 | %(CD8+ESAT6) - %(CD8+ Unstim |
| Tertiary | sin IFNγ (WB) | Ag85 | %(CD8+ Ag85) - %(CD8+ Unstim) |
| Tertiary | sin IFNγ (WB) | Rv2660c | %(CD8+ RV2660c) – %(CD8+ Unstim) |
| Tertiary | sin_IFNγ (WB) | PPD | %(CD8+ PPD) - %(CD8+ Unstim) |
| Tertiary | sin IL2 (WB) | ESAT6 | %(CD8+ ESAT6) - %(CD8+ Unstim) |
| Tertiary | sin_IL2 (WB) | Ag85 | %(CD8+ Ag85) - %(CD8+ Unstim) |
| Tertiary | sin_IL2 (WB) | Rv2660c | %(CD8+ RV2660c) - %(CD8+ Unstim) |


<sup>\*</sup>All samples with an invalid positive control will be excluded from analyses. Invalid positive control is defined as: Invalid if SEB induced tot\_IFNy response by CD4 is < 4 Medians of the tot\_IFNy response by CD4 T cells of the unstimulated controls of all participants in the study at the respective measurement time point.

| Tertlary sin_IL2 (WB) PPD %(CD8+ IPSD) - %(CD8+ Instim) | | (14/5) | DDD | 9/ (CD9 + DDD) 9/ (CD9+ Unctim) |
|---|---|---|---|---|
| Tertiary Sin_TNFa (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) | · | | | |
| Tertiary sin_TNFa (WB) PPD %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary sin_TNFa (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_IFNy/IL2 (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary duo_IFNy/IL2 (WB) Ag85 %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/IL2 (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/INFa (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) ESAT6 %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) Ag85 %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) PPD %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) PPD %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) Ag85 %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) Ag85 %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) PPD %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) PPD %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) PPD %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNy (WB) ESAT6 %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNy (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNy (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNy (WB) PPD %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNy (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNY (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNY (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNY (WB) RV2660c %(CD8+ RV2660c) - %(CD8+ Unstim) Tertiary to_IFNY (WB) RV2660c %(CD8+ | • | | | |
| Tertiary sin_TNFa (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) | - | <del>_</del> | _ | |
| Tertiary duo_IFNy/IL2 (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) | · | <del>-</del> | | |
| Tertiary duo_FNy/IL2 (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary duo_FNy/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_FNy/IL2 (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_FNy/INFa (WB) ESAT6 %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_FNy/TNFa (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary duo_FNy/TNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) PPD %(CD8+ Unstim) Tertiary tot_IFNy (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFN (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim | | | | |
| Tertiary duo_IFNy/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/IL2 (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFa (WB) ESAT6 %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) PPD %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_TNFa/IL2 (WB) PPD %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFa (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) ESAT6 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ BSAT6) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ BSAT6) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_ITNFa (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_ITNFa (WB) Rv2660c %(CD8+ Rv2660c) - | • | | | · · |
| Tertiary duo_ FNy/IL2 (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) | | _ , , , | - | • |
| Tertiary duo_IFNy/TNFα (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) | • | <b>-</b> ' ' ' | | |
| Tertiary duo_ FNy/TNFα (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) | - | | | |
| Tertiary duo_IFNy/TNFα (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_IFNy/TNFα (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_TNFα/IL2 (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary duo_TNFα/IL2 (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary duo_TNFα/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary duo_TNFα/IL2 (WB) PPD %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) ESAT6 %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_INFα (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_INFα (WB) Rv2660c %(CD8+ Ry2660c) - %(CD8+ Unstim) Tertiary tot_INFα (WB) Rv2660c %( | Tertiary | | | , |
| Tertiary duo_IFNy/TNFα (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary duo_TNFα/IL2 (WB) | Tertiary | _ | | - / |
| Tertiary duo_TNFα/IL2 (WB) Ag85 %(CD8+ ESAT6) – %(CD8+ Unstim) | Tertiary | duo_IFNγ/TNFα (WB) | | |
| Tertiary | Tertiary | duo_IFNγ/TNFα (WB) | PPD | |
| Tertiary duo_TNFa/IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) | Tertiary | duo_TNFα/IL2 (WB) | ESAT6 | |
| Tertiary duo_TNFc/IL2 (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) ESAT6 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) Ag85 %(CD8+ Ag85) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IFNY (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNY (WB) PPD %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_IFNY (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ ESAT6) - %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ Rv2660c) - %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ PPD) - %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 % | Tertiary | duo_TNFα/IL2 (WB) | Ag85 | |
| Tertiary tri_IFNy/IL2/TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim Tertiary tri_IFNy/IL2/TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ | Tertiary | duo_TNFα/IL2 (WB) | Rv2660c | |
| Tertiary tri_IFNy/IL2/TNFα (WB) Ag85 | Tertiary | duo_TNFα/IL2 (WB) | PPD | %(CD8+ PPD) - %(CD8+ Unstim) |
| Tertiary tri_IFNy/IL2/TNFα (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tri_IFNy/IL2/TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_INFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Secondary All_Cytokine WB Ag85b SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | $tri_IFN\gamma/IL2/TNF\alpha$ (WB) | ESAT6 | %(CD8+ ESAT6) - %(CD8+ Unstim |
| Tertiary tri_IFNy/IL2/TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) PPD %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ Rv2660c) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, | Tertiary | $tri_IFN\gamma/IL2/TNF\alpha$ (WB) | Ag85 | %(CD8+ Ag85) - %(CD8+ Unstim) |
| Tertiary tot_IFNy (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2 | Tertiary | tri_IFN $\gamma$ /IL2/TNF $\alpha$ (WB) | Rv2660c | %(CD8+ RV2660c) - %(CD8+ Unstim) |
| Tertiary tot_IFNγ (WB) | Tertiary | $tri_IFN\gamma/IL2/TNF\alpha$ (WB) | PPD | %(CD8+ PPD) - %(CD8+ Unstim) |
| Tertiary tot_IFNy (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IFNy (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_INFα (WB) ESAT6 %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Ag85b SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Sun of | Tertiary | tot_IFNγ (WB) | ESAT6 | %(CD8+ ESAT6) - %(CD8+ Unstim) |
| Tertiary tot_IFNγ (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ RV2660c) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Ag85b SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary | Tertiary | tot_IFNγ (WB) | Ag85 | %(CD8+ Ag85) - %(CD8+ Unstim) |
| Tertiary tot_IL2 (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Ag85b SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Sun_TNFα) for PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_IFNγ (WB) | Rv2660c | %(CD8+ RV2660c) - %(CD8+ Unstim) |
| Tertiary tot_IL2 (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB PPD SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_IFNγ (WB) | PPD | %(CD8+ PPD) - %(CD8+ Unstim) |
| Tertiary tot_IL2 (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Ag85b SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_IL2 (WB) | ESAT6 | %(CD8+ ESAT6) - %(CD8+ Unstim) |
| Tertiary tot_IL2 (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB PPD SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_IL2 (WB) | Ag85 | %(CD8+ Ag85) - %(CD8+ Unstim) |
| Tertiary tot_TNFα (WB) ESAT6 %(CD8+ ESAT6) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_IL2 (WB) | Rv2660c | %(CD8+ RV2660c) - %(CD8+ Unstim) |
| Tertiary tot_TNFα (WB) Ag85 %(CD8+ Ag85) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Ag85b SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB PPD SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Sum of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Sum of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Sum of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Sum of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_IL2 (WB) | PPD | %(CD8+ PPD) - %(CD8+ Unstim) |
| Tertiary tot_TNFα (WB) Rv2660c %(CD8+ RV2660c) – %(CD8+ Unstim) Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) – %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Ag85b SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_TNFα (WB) | ESAT6 | %(CD8+ ESAT6) - %(CD8+ Unstim) |
| Tertiary tot_TNFα (WB) PPD %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Ag85b SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_TNFα (WB) | Ag85 | %(CD8+ Ag85) - %(CD8+ Unstim) |
| Tertiary tot_TNFα (WB) PPD %(CD8+ PPD) - %(CD8+ Unstim) Secondary All_Cytokine WB ESAT6 Secondary All_Cytokine WB Ag85b Secondary All_Cytokine WB Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Sum of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Sum of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | Tertiary | tot_TNFα (WB) | Rv2660c | %(CD8+ RV2660c) - %(CD8+ Unstim) |
| Secondary All_Cytokine WB ESAT6 SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for ESAT6 Secondary All_Cytokine WB Ag85b SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Ag85 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | • | tot_TNFα (WB) | PPD | %(CD8+ PPD) - %(CD8+ Unstim) |
| Secondary All_Cytokine WB Ag85b sin_TNFα) for Ag85 Secondary All_Cytokine WB Rv2660c SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for Rv2660c Secondary All_Cytokine WB PPD SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD Secondary All_Cytokine WB SUM (ESAT6+ SUM of (tot_IFNy, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD | | All_Cytokine WB | ESAT6 | sin_TNFa) for ESAT6 |
| Secondary All_Cytokine WB RV2660C sin_TNFα) for Rv2660C Secondary All_Cytokine WB PPD sum (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin_TNFα) for PPD SUM (ESAT6+ SUM of (tot_IFNγ, duo_IL2/TNFα, sin_IL2, sin | Secondary | All_Cytokine WB | Ag85b | sin_TNFa) for Ag85 |
| Secondary All_Cytokine WB PPD sin_TNFα) for PPD sin_TNFα, sin_IL2, | Secondary | All_Cytokine WB | Rv2660c | sin_TNFα) for Rv2660c |
| Consendent All Cytokino MB | Secondary | All_Cytokine WB | | sin_TNFα) for PPD |
| | Secondary | All_Cytokine WB | | |


| Tertiary | tri IFNγ/IL2/TNFα (WB) | SUM (ESAT6+ | SUM of (tri_IFNγ/IL2/TNFα) for ESAT6, |
|---|---|---|---|
| 1 Citial y | ai_ii (4/162/1/4 & (4/2) | Ag85+Rv2660c) | Ag85 and Rv2660c |
| T = .41 = .= . | due IENVII 2 (MD) | SUM (ESAT6+ | SUM of (duo_IFNy/IL2) for ESAT6, Ag85 |
| Tertiary | duo_IFNγ/IL2 (WB) | Ag85+Rv2660c) | and Rv2660c |
| | L. JENL THE - (MID) | SUM (ESAT6+ | SUM of (duo_IFNγ/TNFα) for ESAT6, Ag85 |
| Tertiary | duo_IFNγ/TNFα (WB) | Ag85+Rv2660c) | and Rv2660c |
| | L U O(TNE (IAID) | SUM (ESAT6+ | SUM of (duo_IL2/ TNFα) for ESAT6, Ag85 |
| Tertiary | duo_IL2/TNFα (WB) | Ag85+Rv2660c) | and Rv2660c |

Colour code: blue=secondary priority; red=primary priority; white=tertiary priority.

Table 9: Definition of outcomes from serology: IgG responses to H56:IC31 protein

| Outcome priority group | Outcome | |
|------------------------|------------------------------------|---|
| Tertiary Hypothesis 1 | IgG antibody responses to H56:IC31 | H |
| Primary Hypothesis 2 | IgG antibody responses to H56:IC31 | |
| Primary Hypothesis 3 | IgG antibody responses to H56:IC31 | |

Colour code: blue=secondary priority; red=primary priority; white=tertiary priority.

#### 5.1.1.4 Pharmacokinetics

Pharmacokintetics of etoricoxib will be measured for selected patients during the first 7-10 days with subsequent measurement of etoricoxib in plasma for patients included in arm 1 and arm 4 at day 14 and day 84. Results will be shown in a Supplementary table.

#### 5.1.1.5. Concomitant medication

Will be summarised and displayed by term and ATC code for each treatment arm and shown in a Supplementary table of individual study participants including co-morbidities, medical history, symptoms, reason for stopping intervention etc.

# The following parameters will be described only in the Clinical Study Report

- Clinical chemistry: Sodium (Na), Potassium (K), Calcium (Ca), Creatinine, Creatinine kinase (CK), ASAT, ALAT, Lactate dehydrogenase (LD), Bilirubin, Amylase, GGT, Cholesterol, glucose, HbA1c, Uric acid,
- Haematology: Whole blood count (WBC), monocytes, lymphocytes, Platelets.
- Vital signs: Respiratory rate, heart rate, systolic blood pressure, diastolic blood pressure.

### **5.1.2 Primary Outcome Definition**

The primary outcome is the occurrence of adverse events (AEs), serious adverse events (SAEs), and suspected unexpected serious adverse reactions (SUSARs) for the following time intervals:

a. Day 0 to day 84 (or date of first vaccination if applicable).

Version Number: 1.0 Corina Rueegg 
Version Date: 16.03.2020 Oslo University Hospital

<sup>\*</sup>All samples with an invalid positive control will be excluded from analyses. Invalid positive control is defined as: Invalid if SEB induced tot\_IFNy response by CD4 cells is < 4 Medians of the tot\_IFNy response by CD4 T cells of the unstimulated controls of all participants in the study at the respective measurement time point.

- b. Day 85 (or date of first vaccination if applicable) to day 154 (or 14 days after last vaccination/last Arcoxia treatment, if applicable).
- c. Day 155 (or 15 days after last vaccination/last Arcoxia treatment, if applicable) to day 238.

If the second vaccination is missing, day 154 is defined as 70 days after the date of day 84.

**AEs** are defined as any unintended sign, symptom or disease in a participant receiving the treatment and which does not necessarily have to be causally related with the treatment. The AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA 22).

SAEs are defined as a medical occurrence that results in death, is life-threatening, requires in-patient hospitalisation or prolongation of the existing hospitalisation, results in disabilities, is a congenital abnormality of birth defect, or requires medical intervention to prevent the outcomes mentioned above. If there is a doubt about an AE being serious or not, it is considered serious.

SUSARs are defined as SAEs that are unexpected as defined in the study protocol (V6\_121016), Section 8.1 and 8.2, pages 32-34 and possibly related to the study treatment.

### 5.1.3 Secondary Outcomes Definitions

All secondary outcomes are listed and defined in the Tables 6 to 9 (Section 5.1 Outcome Definitions).

### 5.1.4 Overview of Outcomes

Table 10. Overview of outcomes analysed in this SAP

| Nr | Level | Outcome | Timeframe | Туре |
|---|---|---|---|---|
| 1 | Primary | Number of AEs, SAEs, and SUSARs | Day 0-84, 85-<br>154 and 155-<br>238 | Counts |
| 2 | Secondary,<br>Hypothesis 1,<br>Priority 1 | Immunogenicity outcomes of primary priority in Table 1 | Day 0-238 | Continuous |
| 3 | Secondary,<br>Hypothesis 2,<br>Priority 1 | Immunogenicity outcomes of primary priority in Table 2 | Day 0-238 | Continuous |
| 4 | Secondary,<br>Hypothesis 3,<br>Priority 1 | Immunogenicity outcomes of primary priority in Table 3 | Day 0-238 | Continuous |
| 5 | Secondary,<br>Hypothesis 1,<br>Priority 2 | Immunogenicity outcomes of secondary priority in Table 1 | Day 0-238 | Continuous |
| 6 | Secondary,<br>Hypothesis 2,<br>Priority 2 | Immunogenicity outcomes of secondary priority in Table 2 | Day 0-238 | Continuous |


| 7 | Secondary,<br>Hypothesis 3,<br>Priority 2 | Immunogenicity outcomes of secondary priority in Table 3 | Day 0-238 | Continuous |
|---|---|---|---|---|
| 8 | Secondary,<br>Hypothesis 1<br>to 3, Priority 3 | Immunogenicity outcomes of tertiary priority in Tables 6-9 | Day 0-238 | Continuous |

# 5.2 Analysis Methods

Because of the explorative nature of the trial and the low number of subjects included, we will mainly use descriptive statistics to present the results of the trial.

### 5.2.1 Primary outcome (Outcome 1, Table 10)

#### 5.2.1.1 Primary Analysis

We will calculate the numbers and proportions of participants in the Safety Analysis Set that experienced an AE, SAE, and SUSAR (see 3.3 Analysis Populations) by study arm and above defined three time intervals. We will also present the number and proportions of participants with 1, 2, or ≥3 AEs, SAEs, and SUSARs; the number and proportion of participants with any treatment related AE and SAE; and, the number and proportion of participants with an AE/SAE leading to study drug discontinuation in each study arm and above defined three time intervals. No formal statistical testing of differences between the study arms will be performed. Further, we will display the total number of AEs, SAEs, SUSARs, treatment related AEs and SAEs, and AEs/SAEs leading to study drug discontinuation independent of number of participants. In addition, we will describe the absolute, number of participants with and proportion of participants with AE, SAE, SUSAR, severe AEs, and AEs leading to study drug discontinuation by system organ class (SOC) and preferred term (PT), without calculating any p-values.

### 5.2.1.2 Assumption Checks and Alternative Analyses

There will be no assumption checks or alternative analyses

### 5.2.1.3 Missing data

We will assess safety as reported.

### 5.2.1.4 Sensitivity analyses

There will be no sensitivity analyses.

### 5.2.2 Secondary outcomes (Outcomes Tables 6-9)

### 5.2.2.1 Main analysis

The following analyses will be performed for all secondary outcomes described in Tables 6-9 (all continuous variables).

Descriptive analysis (graphical display of the data) in the FAS:


All the outcomes listed in Tables 6-9 will be described as medians with IQRs over each study time point from 0 to 238 (day 0, 84, 98, 140, 154, 238) by ITT study arm.

All the outcomes listed in Tables 6-9 will be described for each individual over each study time point from 0 to 238 (day 0, 84, 98, 140, 154, 238), stratified by ITT study arm.

For the IgG antibody response to H56:IC31 (Table 9) we will describe the proportion of participants with a twofold increase in response from baseline at any time point during the study, stratified by study arm.

Additional descriptive Figures will be made to graphically display the secondary outcomes of primary priority according to the hypothesis stated in Tables 1-3.

# Statistical analysis and hypothesis testing (according to the statistical framework described in section 2.4) in the FAS:

The secondary outcomes of primary priority for hypothesis 1 (Section 2.4.1) are the response to treatment defined as the change from day 0 to day 84 in the defined readouts. The outcomes will be analysed using median regression with treatment as only independent explanatory factor. The treatment difference of the combination of Arm 1 and 4 (treated with a COX-2 inhibitor) and the combination of Arm 2 and 3 (control) will be presented as estimated difference in median response with 95% confidence interval based on 1000 bootstrap replications and corresponding two-sided p-value.

The secondary outcomes of primary priority for hypothesis 2 (Section 2.4.2) and hypothesis 3 (Section2.4.3) are the responses to vaccine treatment defined as the change from day 84 to day 154 in the defined readouts. The outcomes for hypothesis 2 and 3 will be analysed and presented as for hypothesis 1.

The seed for the bootstrap replications will be set to the date of the final statistical analysis plan (Version 1.0), in the format yyyymmdd.

### 5.2.2.2 Assumption Checks and Alternative Analyses

The median regression with bootstrap-estimated standard error and confidence interval is robust to skewed data and with small sample sizes. There will be no alternative analyses.

### 5.2.2.3 Missing Data

Descriptive statistics and hypothesis testing will be based on available data.

#### 5.2.2.4 Sensitivity Analyses

No sensitivity analyses will be performed.

# 6 Safety Analyses

Safety is the primary outcome of this trial and all performed safety analyses are described under 5.2.1 Primary Analysis.

### 7 Statistical Software

All statistical analyses will be done in Stata v16 or newer (StataCorp. 2015. Stata Statistical Software: Release 16.1 College Station, TX, USA).

### 8 References

### 8.1 Literature References

- 1. Gamble C, Krishan A, Stocken D, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. *Jama* 2017; **318**: 2337-43.
- 2. WHO (2018). Global tuberculosis report 2018, L.C.B.-N.-S. IGO., ed. (Geneva: World Health Organization: Geneva: World Health Organization).

# 8.2 Reference to Data Handling Plan

The Data Handling Plan is appended to this SAP in Appendix II.


### APPENDIX I – The CONSORT flow diagram



### **CONSORT 2010 Flow Diagram**



**APPENDIX II – Data Handlings Plan**